CLINICAL TRIAL: NCT05262959
Title: A Single Center Study of Donafenib Combined With Programmed Cell Death-1 （PD-1） + Transarterial Chemoembolization (TACE) in the First-line Treatment of Advanced Hepatocellular Carcinoma (aHCC)
Brief Title: A Single Center Study of Donafenib Combined With PD-1 + TACE in the First-line Treatment of aHCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-631R
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Donafenib
Keywords: Donafenib; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib (Experimental): Donafenib: 0.1g po. BID. And it will be taken on the first day of the study. PD-1: 200mg ivgtt. Q3W. It will be used at the same time as Donafenib. TACE: The first treatment will be carried out 2-3 weeks after taking Donafenib.
  Interventions: Drug: Donafenib, PD-1; Procedure: TACE

INTERVENTIONS:
Drug: Donafenib, PD-1 — Eligible subjects will receive Donafenib combined with PD-1 and TACE. Donafenib will be taken orally twice a day, 0.1mg each time.PD-1 will be used intravenously every 3 weeks.
Procedure: TACE — TACE will be performed by the investigator based on the patient's tumor status.

SUMMARY:
This study is expected to recruit 30 patients with unresectable HCC who will be treated with Donafenib combined with PD-1 + TACE. During the study period, the tumor efficacy and resectability will be evaluated by imaging examination every 6 weeks. Patients with successful transformation can choose hepatectomy or observation. During the study, safety evaluation and effectiveness evaluation will be carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily enter the study and sign informed consent form (ICF);
2. Age ≥ 18 years and ≤ 75 years, and there is no limit on the gender;
3. Clinically or histologically diagnosed as unresectable HCC;
4. There is at least one measurable lesions that meet the mRECIST standard;
5. Child-pugh classification A or B (score≤7);
6. ECOG : 0 ~ 1 ;
7. The number of intrahepatic tumors ≤ 10 and the maximum tumor diameter ≤ 10cm;
8. Previous TACE treatment ≤ 1 time;
9. Life expectancy ≥ 3 months;
10. For patients with HBV infection, if HBV-DNA is≥10^4copies/ml within 14 days before enrollment, they should take antiviral treatment first, reduce 1 log or reduce to <10^4copies/ml before entering the study, and continue antiviral treatment and monitor liver function and serum HBV-DNA levels;
11. Baseline blood routine and biochemical indexes meet the following criteria within 14 days before treatment:

    Blood routine examination criteria must be met: (no blood transfusion within 14 days)
    1. HB≥90g/L；
    2. ANC≥1.5×10^9/L；
    3. PLT≥70×10^9/L.

    Biochemical tests are subject to the following criteria:
    1. BIL <1.25xULN ；
    2. ALT and AST<5xULN；
    3. Serum creatinine. Less than 1.5 times the upper limit of normal value, Endogenous creatinine clearance>50ml/min ( Cockcroft-Gault formula)；
    4. Albumin≥28g/L；
    5. Electrolytes (phosphorus, calcium, magnesium, potassium) ≥ LLN;
    6. Urine protein <2+ or 24-hour urine protein quantitative detection ≤1.0 g/L.

    Blood coagulation indexes are subject to the following criteria:
    1. Prothrombin time (PT) and international normalized ratio (INR) ≤1.5 × ULN;
    2. Activated partial thromboplastin time（APTT）≤1.5 × ULN.
12. The serum pregnancy test results of female patients with fertility (referring to premenopausal or non surgical sterilization) must be negative within 14 days before enrollment.

Exclusion Criteria:

1. Pathologically confirmed hepatocellular carcinoma intrahepatic cholangiocarcinoma (HCC-ICC) mixed or fibrolamellar hepatocellular carcinoma;
2. The presence of a tumor thrombus in the main portal vein, biliary tract tumor thrombus, inferior vena cava tumor thrombus, or extrahepatic metastasis;
3. Hepatocellular carcinoma recurrence within 2 years after radical resection or ablation;
4. History of malignancy other than HCC within 5 years;
5. Esophageal and/or gastric varices bleeding within 4 weeks prior to initiation of study treatment;
6. Presence of uncontrolled hepatic encephalopathy, hepatorenal syndrome, ascites, pleural effusion, or pericardial effusion;
7. Patients who received liver transplant surgery, prior systemic therapy (chemotherapy, targeted therapy or immunotherapy) or palliative local treatment ≥2 times for HCC；
8. History of organ and cell transplantation；
9. TACE contraindications identified by the investigator;
10. Active severe infection;
11. Autoimmune disease or immune deficiency;
12. Severe organ (heart, kidney) dysfunction;
13. Pregnant or breastfeeding women, and women or men with fertility who are unwilling or unable to take effective contraceptive measures;
14. Unable to follow the research protocol for treatment or scheduled follow-up; Any other researcher who thinks they cannot be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival 1(PFS 1) | an average of 1 year
  PFS 1 refers to the time from the date of enrollment to the first documented tumor progression as assessed by mRECIST criteria or death from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) per mRECIST | an average of 1 year
  The proportion of patients exhibiting a complete response or partial response to treatment, as assessed by mRECIST.
Disease control rate (DCR) per mRECIST | an average of 1 year
  The proportion of patients exhibiting a complete response, partial response or stable disease, as assessed by mRECIST.
Overall survival (OS) | an average of 1.5 year
  The time from the date of enrollment to the date of death from any cause.
Adverse events and serious adverse events. | an average of 1.5 year.
  Incidence of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, M.D., Ph.D., Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai, China.; Zhiping Yan, M.D., Ph.D., Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai, China.
Locations (1):
- Zhongshan Hospital, Fudan University,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No